CLINICAL TRIAL: NCT05605236
Title: Stereotactic Margins in Localized Bronchial Cancer (T1/T2a, N0)
Acronym: Stereotactic
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7460
Record Dates: First submitted 2022-10-28; First posted 2022-11-04 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Bronchial Cancer
Keywords: Bronchial cancer; Bronchopulmonary cancer; Stereotactic radiotherapy; Stereotactic CTV margins; Cell lung cancer; 3D radiotherapy
MeSH Terms: conditions — Carcinoma, Bronchogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bronchopulmonary cancer is the first cause of mortality in the world. We want to update the margins used in stereotactic radiotherapy, in the context of localized lung cancer, of non-surgical management.

The investigators wish to redefine the stereotactic radiotherapy margins according to the histological type in localized non-small cell lung cancer.

Indeed, these criteria were previously defined on a smaller cohort, in the context of 3D radiotherapy (mainly T3, T4 tumors). In addition, the incidence of radiation pneumonitis is highly dependent on the irradiated lung volume, which in turn depends on the CTV margins used.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject operated on at HUS for T1/T2a N0 stage lung adenocarcinoma or squamous cell carcinoma before 30/09/2019
* CT scan available on the HUS imaging server or on CD
* Subject who has not expressed opposition to the use of his or her data for research purposes

Exclusion Criteria:

* Subject who has expressed opposition to participating in the study
* Impossibility to give the subject informed information (difficulties in understanding the subject, ...)
* Subject under legal protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) operated on at HUS for T1/T2a N0 stage lung adenocarcinoma or squamous cell carcinoma before 30/09/2019
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-02-16 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-07-16 (Actual)

PRIMARY OUTCOMES:
Retrospective histological study of tumor cell dissemination around the tumor | Files analysed retrospectively from January 01, 2009 to December 31, 2019 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de chirurgie thoracique - CHU de Strasbourg - France, Strasbourg, France